CLINICAL TRIAL: NCT04802486
Title: Evaluating the Effects of a 12 Week Home-based Exercise Intervention on Physical Performance in Patients With Cancers of the Gastrointestinal Tract With Pre- Cachexia or Cachexia: A Pilot Study
Brief Title: The Effects of a 12 Week Home-based Exercise Intervention on Physical Performance in Patients With Cancers of the Gastrointestinal Tract With Pre- Cachexia or Cachexia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Richard Dunne, Assistant Professor - Department of Medicine , Hematology/Oncology, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UGIM16011
Record Dates: First submitted 2021-03-12; First posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Cachexia; Weight Loss; Gastrointestinal Cancer
Keywords: Cachexia; Weight Loss; Exercise; Gastrointestinal Cancer
MeSH Terms: conditions — Cachexia; Weight Loss; Gastrointestinal Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Exercise Intervention and Standard Care (Experimental): A home-based exercise intervention as well as standard care for your cancer as prescribed by your oncologist
  Interventions: Other: EXCAP©®
- Arm 2: Standard Care (No Intervention): Standard care for your cancer as prescribed by your oncologist

INTERVENTIONS:
Other: EXCAP©® — EXCAP©® is a home-based low-to-moderate intensity program that employs a tailored walking prescription and total body resistance exercises
  Arms: Arm 1: Exercise Intervention and Standard Care

SUMMARY:
The main purpose of this research study is to determine if exercise improve or worsen cachexia.

DETAILED DESCRIPTION:
In this study the investigator would like to better understand how cachexia may improve or worsen, and how exercise may impact this process. The investigator would like to see whether a progressive resistance exercise program (EXCAP©®, Exercise for Cancer Patients) can improve symptoms in patients with gastrointestinal cancers with weight loss and cachexia. The investigator would also like to find out if this exercise intervention improves physical performance, day-to-day function, quality of life, and how exercise may affect different markers in the blood over time.

ELIGIBILITY:
Inclusion Criteria:

* Have a primary diagnosis of colorectal, esophageal, gastric, pancreatic or biliary tract cancer and plans to initiate systemic chemotherapy within the next 4 weeks after enrollment.
* Have been diagnosed as having an advanced unresectable cancer with no plans for surgical intervention during the active study period (12 weeks).
* Have an ECOG performance score of 0 or 1.
* Have a life expectancy of >3 months as determined by their primary oncologist.
* Have experienced at least 2% weight loss of the patient's reported previous body weight over the 6 months prior to enrollment. Patients who have 2 - 4.9% weight loss should also have one of the following metabolic changes: a hemoglobin level <13, an albumin level <3.5, and/or impaired glucose tolerance within the past year such as a new diagnosis of diabetes, an A1C level >5.7, a random glucose level >200 or a fasting glucose level >100.
* Have permission from primary oncologist to engage in low to moderate intensity exercise regimen.
* Be able to read English (since the assessment materials are in printed format).
* Be able to give written informed consent.

Exclusion Criteria:

* Have any of the following limitations: unable to walk the 4 meters of the SPPB test, wheel-chair bound, unable to perform low-to-moderate intensity exercise regimen (patients unable to perform 6 minute walk or stair climb test will be allowed to participate, but will be held out of these measurements).
* Have had major surgery (excluding diagnostic procedures like laparoscopy, EGD/EUS, esophageal stent placement) in the past 4 weeks.
* Be experiencing dysphagia that requires enteral or parenteral feeding for nutrition.
* Be enrolled on hospice at time of consent.
* Be engaged in an active exercise routine by being identified as in the Active or Maintenance Stage of exercise behavior as assessed by the 1-item Exercise Stages of Change Short Form (40).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-06-29 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
Number of patients that adhered to the exercise conditions of the study | 3 Months
  Measured by the Short Physical Performance Battery (SPPB) in patients with advanced GI malignancies

SECONDARY OUTCOMES:
Porportion of subjects with improved cachexia-related symptoms 3 months | 3 Months
  The Functional Assessment of Anoreix/Cachexia Therapy subscale is a 39-item questionnaire that measures general aspects of quality of life as well as specific anorexia/cachexia-related concerns. This will be collected at pre- and post intervention

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No